CLINICAL TRIAL: NCT01986751
Title: Effectiveness of Perineural Clonidine as an Adjuvant With Ropivacaine for Popliteal Nerve Block in Patients Undergoing Foot and Ankle Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: failure to enroll
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Promil Kukreja, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F130625002
Record Dates: First submitted 2013-10-31; First posted 2013-11-18 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-07

CONDITIONS: Pain
Keywords: nerve; block; motor blockade; lower extremity pain; nerve block
MeSH Terms: conditions — Pain; Bites and Stings | interventions — Clonidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine and Ropivacaine (Experimental): A bolus of 20 mL of 0.5% ropivacaine mixed with clonidine 1mcg/kg will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose).
  Interventions: Drug: Clonidine; Drug: ropivacaine
- Ropivacaine (Active Comparator): Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: Clonidine
  Other Names: Catapres, Kapvay, Nexiclon, Jenloga, Duraclon
  Arms: Clonidine and Ropivacaine
Drug: ropivacaine

SUMMARY:
Nerve blocks are used to decrease the amount of pain you have after surgery. We are asking you to take part in a research study. This research study will test whether adding a medicine called clonidine to nerve blocks helps to improve them. Nerve blocks typically last less than a day after surgery. We are looking for ways to make them work better and last longer. Clonidine is approved for use as a blood pressure medicine. Its use in nerve blocks is investigational, but it may help nerve blocks to last longer. Adding clonidine to nerve blocks may also decrease the amount of pain medicine a person has after surgery. All people who enter this study will receive a nerve block with the normal medicine, but half of people will also have clonidine added to their nerve block. This study will enroll 60 participants from UAB hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing foot or ankle surgery with popliteal nerve block planned for postoperative analgesia.
2. Adult, 19 years of age and older.
3. Subject classified as American Society of Anesthesiology (ASA) class 1, 2, or 3. The ASA defines these statuses as follows: 1-A normal healthy patient. 2-A patient with mild systemic disease. 3-A patient with severe systemic disease.

   -

Exclusion Criteria:

1. Any subject not classified as an ASA 1, 2, or 3.
2. Allergy/intolerance to local anesthetic, clonidine, and/or oxycodone.
3. Subject with a history of continuous opioid use for greater than one month prior to surgery.
4. Pre-existing neurologic deficit in lower extremity (surgical site).
5. Clinically significant coagulopathy (hemophilia, von Willebrand disease).
6. Patients who fail to follow the UAB Department of Anesthesiology Algorithm for the Preoperative Management of an Angiotensin Converting Enzyme Inhibitor (ACEI) or an Angiotensin Receptor Blocker (ARB). A copy of the algorithm can be found in Appendix 1. -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Promil Kukreja, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clonidine and Ropivacaine: A bolus of 20 mL of 0.5% ropivacaine mixed with clonidine 1mcg/kg will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose).
  Clonidine
  ropivacaine
- Ropivacaine: Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine
  ropivacaine
Period: Overall Study
Arm/Group | Clonidine and Ropivacaine | Ropivacaine
Started | 10 | 4
Completed | 0 | 2
Not Completed | 10 | 2
Not completed — improperly consented | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine and Ropivacaine | Ropivacaine | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Onset of Sensory and Motor Block Between the Study Group and the Control Group
Description: Mean time onset of sensory block and motor block between the study group and the control group to assess the efficacy of clonidine to prolong the block duration.
Time Frame: baseline to 72 hours
Population: Study was prematurely terminated. No data were collected for this assessment.
Groups:
- Clonidine and Ropivacaine (Study Group): A bolus of 20ml of 0.5% ropivacaine mixed with clonidine 1mcg/kg will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose).Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine.
- Ropivacaine (Control): A bolus of 20ml of 0.5% ropivacaine will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose).Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine.
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Compare the Mean Duration of Sensory and/or Motor Block Between the Study Group and the Control Group
Description: Mean duration of sensory and/or motor block between the study group and the control group to assess the efficacy of clonidine to prolong the block duration.
Time Frame: baseline to 72 hours
Population: Study was prematurely terminated. No data were collected for this assessment
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Compare the Mean VAS Scores at 24 Hours Post Procecure to Determine the Effectiveness of Perineural Clonidine on Duration of Postoperative Analgesia Between the Control Group and Study Group
Description: The VAS score is measured as 0 - 10 with 0 being no pain to 10 being the worst pain imaginable to assess the efficacy of clonidine to control postoperative pain and patient satisfaction at the time of discharge.
Time Frame: baseline to 24 hours post block
Population: Study was prematurely terminated. No data were collected for this assessment
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Compare the Opioid Consumption During the First 24 Hours Between the Study Group and the Control Group
Description: Mg equivalent of morphine consumption during the first 24 hours between the study group and the control group
Time Frame: baseline to 24 hours post block
Population: Study was prematurely terminated. No data were collected for this assessment
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Compare the Subjects Mean Arterial Blood Pressure Effect of Perineural Clonidine Versus Placebo
Description: Comparing the mean arterial blood pressure between the study group and the control group to assess the effect of clonidine on blood pressure.
Time Frame: baseline to discharge from hospital (expected 3 days)
Population: Study was prematurely terminated. No data were collected for this assessment
Groups:
- Clonidine and Ropivacaine (Study Group): A bolus of 20ml of 0.5% ropivacaine mixed with clonidine 1mcg/kg will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose). Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine.
- Ropivacaine (Control): A bolus of 20ml of 0.5% ropivacaine will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose). Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine.
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: the Mean Time to Discharge After Start of Procedure for Each Group - Control and Study Group.
Description: Comparing the mean hours from start of procedure to discharge between the study group and the control group
Time Frame: baseline to discharge (approximately 72 hours)
Population: Study was prematurely terminated. No data were collected for this assessment
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Time to First Analgesic Intake Postoperative Between the Control Group and the Study Group.
Description: Comparing the mean time to the first analgesic intake postoperative between the control group and the study group
Time Frame: baseline to 24 hours post block
Population: Study was prematurely terminated. No data were collected for this assessment
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Compare the Mean VAS Scores at 24 Hours Post Procedure to Determine the Patient Satisfaction on Duration of Postoperative Analgesia Between Control Group and Study Group
Description: Compare the mean VAS scores at 24 hours between the study group and the control group to assess the efficacy of clonidine to control postoperative pain and patient satisfaction at the time of discharge.
Time Frame: baseline to 24 hours
Population: Study was prematurely terminated. No data were collected for this assessment
Groups:
- Clonidine and Ropivacaine: A bolus of 20ml of 0.5% ropivacaine mixed with clonidine 1mcg/kg will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose). Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine.
- Ropivacaine: A bolus of 20ml of 0.5% ropivacaine will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose). Standard saphenous nerve block (adductor canal approach) will be performed using 15ml of 0.5% ropivacaine.
Arm/Group | Clonidine and Ropivacaine | Ropivacaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Clonidine and Ropivacaine (Study Group): A bolus of 20 mL of 0.5% ropivacaine mixed with clonidine 1mcg/kg will be injected through the stimulating needle with gentle aspiration between divided doses (5 mL per dose).
- Ropivacaine (Control): Standard saphenous nerve block (adductor canal approach) will be performed using 20 ml of 0.5% ropivacaine
Arm/Group | Clonidine and Ropivacaine (Study Group) | Ropivacaine (Control)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 0/10 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No